CLINICAL TRIAL: NCT02109900
Title: Prognostic Value of Progesterone Levels on Oocyte Retrieval Day for Outcome of Intracytoplasmic Sperm Injection
Brief Title: Prognostic Value of Progesterone on Oocyte Retrieval Day for In Vitro Fertilization Outcome
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Turgut Aydın, Specialist, Gynecology and Obstetrics, Acibadem University
Other Study IDs: OpudayPivfOutcome
Record Dates: First submitted 2014-04-07; First posted 2014-04-10 (Estimated); Last update posted 2014-04-10 (Estimated); Status verified 2014-04

CONDITIONS: Infertility; Assisted Reproductive Technology
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Serum Progesteron Levels
  Interventions: Other: Serum Progesterone Levels

INTERVENTIONS:
Other: Serum Progesterone Levels

SUMMARY:
This observational study aims the potential role of serum progesterone levels on the day of oocyte pick-up on the probability of pregnancy, in patients undergoing antagonist IVF cycles.

There has been evidence, that increased serum levels of progesterone on triggering day are associated with a decreased probability of pregnancy after IVF.

There is no study that investigate assocation between serum progesterone levels on the day of oocyte pick-up and IVF outcomes. This study will be the first in this case.

ELIGIBILITY:
Inclusion Criteria:

* Age < 40 years
* Basal FSH < 12 IU/L
* Basal P < 1.6 ng/mL

Exclusion Criteria:

* Women with polycystic ovaries syndrome (PCOS)
* Women with Stage III-IV Endometriosis
* Women with a pathological condition of the adrenal glands

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients who are referred to Acibadem Kayseri Hospital IVF Unit
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2014-02; Primary Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy | At 6-8 weeks of gestation
  Clinical pregnancy, defined as ultrasound evidence of gestational sac at 6 weeks of gestation

CONTACTS AND LOCATIONS:
Overall Officials: Turgut Aydin, Principal Investigator — Acıbadem Kayseri Hospital